CLINICAL TRIAL: NCT02002260
Title: Levonorgestrel Intrauterine System Versus Oral Contraceptives for Heavy Menses
Brief Title: Stopping Heavy Periods Project
Acronym: SHiPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Kristen Matteson , M.D., Associate Professor of Obstetrics and Gynecology, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HD074751 (NIH)
Record Dates: First submitted 2013-11-27; First posted 2013-12-05 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Abnormal Uterine Bleeding; Abnormal Uterine Bleeding, Ovulatory Dysfunction; Abnormal Uterine Bleeding, Endometrial Hemostatic Dysfunction
MeSH Terms: conditions — Metrorrhagia | interventions — Contraceptives, Oral, Combined; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levonorgestrel intrauterine system (Active Comparator): levonorgestrel intrauterine system with 52 mg of levonorgestrel, levonorgestrel is released at a rate of approximately 20 μg/day. Inserted once, duration 5 years.
  Interventions: Device: Levonorgestrel intrauterine system
- Combined oral contraceptives (Active Comparator): A combined ethinyl estradiol (ee) and progestin oral contraceptive pill chosen by the participants' primary gynecologic care provider. Monophasic with 30 or 35 mcg ee administered according to pill pack instructions (21 days active pills, 7 placebo pills)
  Interventions: Drug: Combined oral contraceptives

INTERVENTIONS:
Device: Levonorgestrel intrauterine system
  Other Names: Mirena
  Arms: Levonorgestrel intrauterine system
Drug: Combined oral contraceptives
  Other Names: Any combined oral contraceptive of the provider's choice so long; as it contains 30-35 mg of ethinyl estradiol.
  Arms: Combined oral contraceptives

SUMMARY:
This study is a randomized clinical trial comparing the effectiveness of the levonorgestrel intrauterine system (LNG-IUS) to combined oral contraceptives (COCs) for improving quality of life among women who report heavy menstrual bleeding.

DETAILED DESCRIPTION:
This study is designed to be conducted within the context of a patient's standard/usual/typical care from their primary gynecologic care provider. We hypothesize that, compared to COCs, the LNG-IUS will be more effective at improving bleeding-related quality of life at 6 months and one year. To test this hypothesis, we plan to enroll 59 women from several sites who present for gynecologic care and self-report heavy menstrual bleeding into a RCT comparing LNG-IUS to COCs. The eligible study population includes women with heavy menstrual bleeding secondary to ovulatory disorders (AUB-O) or endometrial hemostatic disorders (AUB-E). Women meeting study eligibility will be randomized to receive LNG-IUS or COCs. Main study outcomes will be obtained at 6 weeks, 3 months, 6 months, and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported heavy menstrual bleeding
* Age 18-51 years
* Etiology of heavy menstrual bleeding from either ovulatory disorders (AUB-O) or endometrial hemostatic disorders (AUB-E)

Exclusion Criteria:

* Plan pregnancy in the next year
* Menopausal
* Currently has a copper IUD in place
* History of ablation or hysterectomy or have any contraindications to COCs or LNG-IUS

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Menstrual Bleeding Questionnaire | Completed 5 times over a one year time period
  We will measure bleeding-specific quality of life using the Menstrual Bleeding Questionnaire (MBQ), a validated tool to assess bleeding-related quality of life, which is the most important outcome for patients and for clinicians treating this symptom. We will measure MBQ score at randomization, and at 6 weeks, 3 month, 6 months, and 12 months post-randomization for both groups

SECONDARY OUTCOMES:
Treatment Failure | Information collected at four time points during a one year period post randomization
  The goal of treating heavy menstrual bleeding is to utilize a treatment option that improves patient quality of life and avoids surgical intervention. We will look at treatment failure two different ways. We will determine the overall proportion of participants who discontinued their assigned treatment (opted for no treatment or chose a different treatment option, including surgery) and subset that opted for surgical intervention (endometrial ablation or hysterectomy) during the study period. This information will be recorded by the primary gynecologic provider (physical examination and physician form), by participants (interval health history form), and by the research team (medical record review).

CONTACTS AND LOCATIONS:
Overall Officials: Kristen A Matteson, M.D., M.P.H., Principal Investigator — Women and Infants Hospital
Locations (1):
- Gynecologic practices affiliated with Women and Infants Hospital, Providence, Rhode Island, United States